CLINICAL TRIAL: NCT05128383
Title: An Open-label Proof of Concept Study Regarding the Efficacy and Safety of Dupilumab in the Treatment of Keloids
Brief Title: Study to Assess Efficacy and Safety of Dupilumab in the Treatment of Keloids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Martina Porter, MD, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000648
Record Dates: First submitted 2021-10-26; First posted 2021-11-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Keloid
Keywords: keloid; keloid scar; hypertrophic scar; scar
MeSH Terms: conditions — Keloid; Cicatrix, Hypertrophic; Cicatrix | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dupilumab Subcutaneous Injection (Experimental): 600 mg at initial visit and 300mg every 2 weeks until week 22
  Each subject will receive 600mg of Dupilumab at baseline visit and 300mg of Dupilumab as a subcutaneous injection every 2 weeks for a total of 9 doses over 22 weeks.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Dupilumab a human monoclonal antibody of the immunoglobulin G4 subclass that inhibits interleukin (IL)-4 and IL-13 signaling by specifically binding to the IL-4 receptor alpha subunit, which is shared by the IL-4 and IL-13 receptor complexes.
  Other Names: Dupixent

SUMMARY:
The study investigates the efficacy and safety of dupilumab in the treatment of keloids

DETAILED DESCRIPTION:
Current scar treatments have limited efficacy and are often unsatisfactory although over $20 billion dollars are spent annually on the treatment and management of scars. Keloids, an abnormal proliferation of scar tissue, can be disfiguring, functionally impairing, and have dramatic impacts on quality of life. Treatments of keloids include a variety of modalities (i.e. intralesional steroid injections, silicone gel or sheets, surgery, laser, radiation therapy, cryotherapy, topical imiquimod, and intralesional 5-fluorouracil injections). However, current treatments are limited to primarily localized interventions.

The Investigators hypothesize that dupilumab can decrease the size and symptoms of keloids and improve patient's quality of life. An open-label proof of concept study regarding the use of dupilumab in patients with keloids may be the first step in elucidating a novel systematic approach to treatment of keloids.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 65 at the time of dupilumab initiation.
* Subjects must have either one keloid with ≥ 2 cm length-wise or at least two keloids with ≥ 0.4 cm (width) x 0.4 cm (length)
* Subjects must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study related activity is performed.

Exclusion Criteria:

* History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis (Tb) infection as defined by a positive QuantiFERON TB-Gold test at screening.
* Known infection with HIV, hepatitis B or hepatitis C at screening.
* Are currently pregnant, breastfeeding, or planning to get pregnant during the study.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unwilling to use effective contraception during the study and for 8 weeks after stopping treatment. Methods of acceptable birth control are listed below under "Women of Childbearing Potential"
* Previous hypersensitivity reaction to dupilumab.
* Patients with acute asthma, acute bronchospasm or status asthmaticus.
* Patients with known helminth infections.
* Currently on any other immunosuppressant systemic medication or within 28 days of baseline visit.
* Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) which in the opinion of the investigator significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy.
* Are participating in another study using an investigational agent or procedure during participation in this study or within 28 days prior to baseline visit.
* Any other treatment for keloids with 28 days prior to baseline visit, including silicone gel/sheets, laser therapy, intralesional steroid or 5-fluorouracil injections, topical steroid, cryotherapy, surgery, or radiation therapy.
* Has had a live vaccine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | Baseline and Week 24
  Average patient scores for Patient and Observer Scar Assessment Scale (POSAS) from baseline and week 24.
  The POSAS measures scar quality by evaluating visual (e.g. color), tactile (e.g. pliability) and sensory (e.g. itch) characteristics of the scar from the perspective of the observer (investigator) and patients. POSAS is comprised of two numeric scales: the Patient Scar Assessment Scale (PSAS, patient scale measuring pain, pruritus, color, stiffness, thickness, bumpiness) and the Observer Scar Assessment Scale (OSAS, observer scale measuring vascularity, pigmentation, thickness, relief, pliability, surface area). Both scales contain six items that are scored numerically on a 1-10 scale. A score of "1" being "no, not at all" and a score of "10" being "yes, very much". Together, they make up the total score (range of 12-120) of the PSAS (range of 6-60) and OSAS (range of 6-60).

SECONDARY OUTCOMES:
Vancouver Scar Scale (VSS). | Baseline and Week 24
  Average score of patients for Vancouver Scar Scale (VSS) from baseline and week 24.
  Score Description:
  The VSS measures four parameters of scars: vascularity, pigmentation, pliability, and height. Each parameter contained ranked subscales that may be summed to obtain a total score ranging from 0 (representing normal skin) to 13 (representing worst scar imaginable).
  * Vascularity: assessed by looking at the scar at resting and by blanching the scar and observing the rate and amount of blood return
    1. Score 0: normal color and capillary refill
    2. Score 1: pink scar with a slight increase in the local blood supply
    3. Score 2: red scar with a significant increase in the local blood supply
    4. Score 3: purple scar with excess local blood supply, scars which are congested and refill slowly or cannot be completely blanched
  * Pigmentation: The skin will be blanched with a piece of plastic to eliminate the effect of vascularity on skin color and compared with normal skin (Score: 0-3)
Dermatology Life Quality Index (DLQI). | Baseline and Week 24
  Average score patient-reported outcomes based on Dermatology Life Quality Index (DLQI).
  Score Description:
  A Quality of Life Score will be calculated based upon the Dermatology Life Quality Index (DLQI).
  The DLQI is a validated general dermatology questionnaire that consists of 10 items that assess subject health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment) (Appendix 3)12. It has been extensively used in dermatology clinical trials for atopic dermatitis. The DLQI is a psychometrically valid and reliable instrument that has been translated into several languages, and the DLQI total scores have been shown to be responsive to change. The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline.
Histology | Baseline and Week 24
  Histology Description:
  Percentage Intensity of expression of the markers will be measured by an image analysis program for patients who have data for both baseline and week 24.
Number of patients with keloid volume and size improvement | Baseline and Week 24
  keloid volume and size improvement will be assessed based on photographs taken by Canfield camera analysis software for patients who have data for both baseline and week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Porter, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No